CLINICAL TRIAL: NCT05783024
Title: ADAM Substudy Luik 2: Observational Retrospective Single Centre Cohort Study on Constructing & Validating AI Prediction Models for Outcomes of Lung Cancer Patients
Brief Title: Advanced Data-Aided Medicine Part Lung Cancer
Acronym: ADAMpartlung
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AZ Delta (Other)
Responsible Party: Sponsor
Other Study IDs: B1172021000032
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer
Keywords: AI; ML; Lung Cancer; Prediction
MeSH Terms: conditions — Lung Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — retrospective data collection

SUMMARY:
Developing and validating an AI model that supports physicians in their decision process for treating lung cancer patients. This AI model needs to predict the probability of (the evolution of) the outcomes, based on clinical data and a simulated lung cancer treatment plan. The outcome probabilities can be evaluated with different treatment plans to identify the optimal plan. Initially, the input data will be a limited set of selected features such as general patient information, tumour characteristics, laboratory measurement results, comorbidities and treatments. Finally, the goal is to use a deep patient as input to the models.This deep patient is an AI model on its own, trained on hospital data, as described in secondary objectives.

DETAILED DESCRIPTION:
The aim of this study is to prepare and unlock siloed real-world-data (RWD) for analysis and artificial model construction with the goal to derive real-world-evidence (RWE). Nowadays physicians and nurses are gathering data from patients and register the data in the electronic health record system. Datapoints are often not available in a structured format, so data gathering and unlocking is done manually upon request. Careful analysis of the collected data using artificial intelligence tools might also help to predict which patients are at the highest risk of unscheduled health care use, emergency department visits and hospital admissions. Therefore, a model able to predict the relevant outcomes would be of significant help to the physicians' daily practice.

Primary Objective Developing and validating an AI model that supports physicians in their decision process for treating lung cancer patients. This AI model needs to predict the probability (of the evolution) of the outcomes, based on clinical data and a simulated lung cancer treatment plan and later on a deep patient. Model input data sources are hospital data like demographics, baseline health status, prior treatments, tumour characteristics, comorbidities , imaging data & physiological data, detailed treatment data.

Secondary Objectives

* Automatic unlocking, collection & transformation of lung cancer datapoints to OMOP common data model so that data is readily available for further research & analysis
* Training and validating supervised machine learning models with a limited feature set as input to predict lung cancer patient outcomes
* Constructing a digital patient by training an AI model fed with all data available in OMOP common data model
* Validating a digital patient & optimal feature selection to enhance AI model performance via unsupervised learning techniques

The potential of applying transformers to represent patients is truly personalized and even predictive medicine. The reason is that transformers are an instrument which make it possible to deal with millions of interacting and non-linearly behaving parameters. Hence data sources can be extended to include genetic information and so on. Optimal feature selection from a digital patient can enhance AI model performance via unsupervised learning techniques, and so further finetune prediction models for daily practice.

To build a virtual twin to represent a patient in detail so population analysis and model building is clinically relevant.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer patients included in the lung cancer patient pathway

Exclusion Criteria:

* None specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lung cancer patients included in the lung cancer patient pathway from 20/04/2018
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2024-09-27 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Data into international common data model ready for AI input | 2022
  Lung cancer hospital data translated and clinically validated in UMLS concepts and stored in the OMOP common data model

SECONDARY OUTCOMES:
Supervised machine learning | 2023
  Training and validating supervised machine learning models with a limited set of selected features as input to predict lung cancer patient outcomes.
Digital patient construction | 2023
  Constructing a digital patient by training an AI model
Construction & validation of predictive AI model for lung cancer patients | 2024
  Construction & validation of predictive AI model feasibility approach; Constructing predicted outcome AI models like 30 day mortality, 30- day ER visit, QoL evolution, acute treatment complications

CONTACTS AND LOCATIONS:
Overall Officials: Ingel Demedts, MD, Principal Investigator — AZ Delta
Locations (1):
- AZ Delta, Roeselare, West-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No